CLINICAL TRIAL: NCT00735059
Title: Test of the Nipro ELISIO H Dialyzer in Different Dialysis Treatment Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EXcorLab GmbH (Other)
Collaborators: Nipro Europe N.V. (Industry)
Responsible Party: Dr. Horst-Dieter Lemke, Biochemist, Chief Executive Officer, EXcorLab GmbH
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KSEL0702
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Last update posted 2009-08-21 (Estimated); Status verified 2009-08

CONDITIONS: Chronic Kidney Disease
Keywords: dialysis membrane; Polynephron; Elisio H; Polyethersulfone; Diapes; PES-DS; online post-dilution hemodiafiltration; hemodialysis; protein-bound toxins; beta-2-microglobulin; hemodialysis patients
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): treatment with dialyzer ELISIO 170H
  Interventions: Device: treatment with the dialyzer ELISIO 170H
- 2 (Active Comparator): treatment with dialyzer PES-170DS
  Interventions: Device: treatment with the dialyzer PES-170DS

INTERVENTIONS:
Device: treatment with the dialyzer ELISIO 170H — one week of three consecutive dialysis treatments, > 3 hours
  Arms: 1
Device: treatment with the dialyzer PES-170DS — one week of three consecutive dialysis treatments, > 3 hours
  Arms: 2

SUMMARY:
A current trend in dialysis membrane engineering is to maximize the permeability for larger low-molecular weight proteins while retaining albumin. Protein-leaking dialysis membranes do not meet these requirements. Particularly in convective procedures, such as hemodiafiltration, their albumin leakage is too high [10]. POLYNEPHRON™, the membrane which is built in to the new Nipro ELISIO® dialyzer, is a new dialysis membrane, produced by applying an innovative spinning technique. The incentive of its development was to improve the characteristics of existing dialysis membranes, i.e., realizing a steeper sieving profile for low-molecular weight proteins without significant loss of essential larger proteins at best biocompatibility properties, for a more adequate dialysis therapy. Purpose of the planned study is to demonstrate the superior performance at lower albumin loss in different dialysis procedures of the new Nipro ELISIO® dialyzer compared with a control dialyzer with regard to the removal of the whole range of uremic toxins.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* CKD stage 5 with hemodialysis or hemodiafiltration treatment for more than three months
* Hematocrit >30 %
* Routine anticoagulation and erythropoietin regimen
* No vascular access related problems (A/V-fistula, graft or bi-flow catheter)
* No ongoing infection
* Signed informed consent form

Exclusion Criteria:

* Inclusion criteria not met
* Known HIV or active hepatitis B or C infection (positive PCR). Pregnancy
* Unstable clinical condition (e.g. cardiac or vascular instability)
* Life expectancy less than 12 months
* Known coagulation problems
* Patients participating in another study interfering with the planned study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
protein-bound toxin removal | pre and post dialysis treatment
low-molecular weight protein removal | pre and post dialysis treatment
small solute removal | pre and post dialysis treatment

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Vanholder, Prof. Dr., Principal Investigator — University Hospital Ghent, Nephrology Section
Locations (1):
- University Hospital, Ghent, Belgium